CLINICAL TRIAL: NCT02468102
Title: A Pharmacoepidemiological Study of Rivaroxaban Use and Potential Adverse Outcomes in Routine Clinical Practice in Sweden
Brief Title: Study of Rivaroxaban Use and Potential Adverse Outcomes in Routine Clinical Practice (Sweden)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 17543; XA1405SE (Other: Company internal)
Record Dates: First submitted 2015-06-08; First posted 2015-06-10 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Acute Coronary Syndrome; Venous Thrombosis; Pulmonary Embolism; Atrial Fibrillation
Keywords: Rivaroxaban; Venous Thrombosis/Pulmonary Embolism; Stroke Prevention in Atrial Fibrillation; Anticoagulants; Hematologic Agents; Therapeutic Uses; Observational; Pulmonary Embolism; Venous Thrombosis; Venous Thromboembolism; Intracranial Hemorrhages; Gastrointestinal Hemorrhage
MeSH Terms: conditions — Acute Coronary Syndrome; Venous Thrombosis; Pulmonary Embolism; Atrial Fibrillation; Venous Thromboembolism; Intracranial Hemorrhages; Gastrointestinal Hemorrhage | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rivaroxaban / Cohort 1: Patients who have filled a prescription for rivaroxaban in any pharmacy in Sweden during the study period.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Standard of care drugs / Cohort 2: Patients who have filled a prescription for standard of care drugs (warfarin, aspirin, clopidogrel, ticlopidine, prasugrel or ticagrelor) in any pharmacy in Sweden during the study period.
  Interventions: Drug: Standard of care drugs

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Treatment of deep vein thrombosis (DVT) or pulmonary embolism (PE), and prevention of recurrent DVT and PE (15 mg rivaroxaban twice daily [bid] for 3 weeks, then 15 mg or 20 mg once daily [od], tablets).
  Prevention of stroke and systemic embolism with non-valvular atrial fibrillation (stroke prevention in atrial fibrillation [SPAF]) with one or more risk factors, prior stroke or transient ischaemic attack (20 mg rivaroxaban [od], tablets).
  Prevention of venous thromboembolism (VTE) in patients undergoing elective hip or knee replacement surgery (recommended dose: 10 mg rivaroxaban [od] tablets for 35 days following hip replacement surgery and 14 days following knee replacement surgery).
  Co-administered with acetylsalicylic acid (ASA) alone or with ASA plus clopidogrel or ticlopidine, for the prevention of atherothrombotic events in patients after an acute coronary syndrome (ACS) with elevated cardiac biomarkers (recommended dose 2.5 mg rivaroxaban tablets [bid]).
  Groups: Rivaroxaban / Cohort 1
Drug: Standard of care drugs — For DVT/PE treatment and SPAF, standard of care is treatment with the most widely used vitamin K antagonist, phenprocoumon, and for the secondary prevention of ACS, standard of care is antiplatelet drug(s) such as low-dose acetylsalicylic acid, clopidogrel, dipyridamole, prasugrel, ticlopidine and ticagrelor.
  Groups: Standard of care drugs / Cohort 2

SUMMARY:
This prospective cohort study will provide information about:

Characteristics of Rivaroxaban use in patients who are prescribed Rivaroxaban for the first time compared to patients who are prescribed standard of care for the first time.

The occurrence of intracranial haemorrhage, gastrointestinal and urogenital bleeding, and the occurrence of non-infective liver disease.

ELIGIBILITY:
Inclusion Criteria:

* All male and female patients who have filled a prescription for rivaroxaban, warfarin, aspirin, clopidogrel, ticlopidine, prasugrel and ticagrelor in any pharmacy in Sweden, between December 9, 2011 and December 31, 2018

Exclusion Criteria:

- For the AF and DVT/PE treatment indications, patients who have filled a prescription for warfarin or another oral anticoagulant at any time between July 1, 2005 and December 9, 2011 will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents of Sweden: The study population will be identified using data from the Swedish national health registers that are maintained by the national Board of Health and Welfare.
Sampling Method: Non-Probability Sample
Enrollment: 99999 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Descriptive analysis of demographic and clinical characteristics of patients who are prescribed oral rivaroxaban for the first time in comparison with those who are prescribed standard of care for the first time | up to 4 years
  The following data will be collected and assessed at 2 and 4 years after rivaroxaban market authorization: • age and sex distribution at index date • dose of rivaroxaban at index date • diagnosis associated with the prescribing of the index drug • use of specific prescribed medications confirming ACS indication • use of other prescribed medications • comorbidity based on diagnoses • renal impairment • healthcare utilization (e.g. outpatient visits and hospital admissions)
Safety and effectiveness: occurrence of hospitalization for a) intracranial haemorrhage, (b) gastrointestinal bleeding, (c) urogenital bleeding among users of rivaroxaban in comparison with individuals receiving current standard of care | up to 5 years
  The two cohorts will be followed up from the index date until 12 months after the end of the enrolment period for potential outcomes For descriptive purposes, annualized crude incidence rates of the major bleeding events will be calculated, accompanied by 95% confidence intervals.
  For evaluation of safety and effectiveness outcome events, Cox proportional hazards regression model will be used. Propensity score matching will be done to account for confounding by indication.

SECONDARY OUTCOMES:
Occurrence of hospitalization for bleeding events not specified as primary safety outcomes ("other bleeding", secondary safety outcome) in individuals receiving rivaroxaban, in comparison with those receiving current standard of care. | at 5 years
  Outcome will be analyzed after end of data collection. Cox proportional hazards regression model will be used. Propensity score matching will be done to account for confounding by indication.
Occurrence of non-infective liver disease (secondary safety outcome) in individuals receiving rivaroxaban in comparison with those receiving current standard of care. | at 5 years
  Outcome will be analyzed after end of data collection. Cox proportional hazards regression model will be used. Propensity score matching will be done to account for confounding by indication.
Outcomes related to effectiveness (DVT/PE, ischaemic stroke or myocardial infarction) in individuals receiving rivaroxaban in comparison with those receiving current standard of care. | at 5 years
  Outcome will be analyzed after end of data collection. Cox proportional hazards regression model will be used. Propensity score matching will be done to account for confounding by indication.
All-cause mortality as well as cause-specific mortality. | at 5 years
  Outcome will be analyzed after end of data collection. Cox proportional hazards regression model will be used. Propensity score matching will be done to account for confounding by indication.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Multiple Locations, Sweden

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/